CLINICAL TRIAL: NCT04161599
Title: Oral + Parenteral Antibiotic Prophylaxis Before Colonic Surgery With vs Without Mechanical Bowel Preparation: a Prospective, Multicentric, Randomised, Controlled Trial.
Brief Title: Preoperative Oral Antibiotics With vs Without Mechanical Bowel Preparation to Reduce Surgical Site Infections Following Colonic Resection: an International Randomized Controlled Trial.
Acronym: ORALEV2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-004283-21
Record Dates: First submitted 2019-11-04; First posted 2019-11-13 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Wounds and Injuries; Surgery--Complications
MeSH Terms: conditions — Wounds and Injuries | interventions — Cefuroxime; Metronidazole; Tablets; picosulfate sodium; Citric Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral + Parenteral prophylaxis + Mechanical Bowel Preparation (Experimental): Drug: Extra dosage - cefuroxime (750mg) I.V
  Procedure: Colonic Surgery Both groups undergo colonic surgery. This section does not include rectal surgery ( see Inclusion/exclusion criteria)
  Drug: Cefuroxime 750mg oral An oral antibiotic pattern of ciprofloxacin (750mg / 12h, 2 doses) the day before surgery.
  Drug: Metronidazole 250mg oral An oral antibiotic pattern of metronidazole (250mg / 8h, 3 doses) the day before surgery.
  Drug: Sodium picosulfate, magnesium oxide, citric acid anhydrous 15.08 g oral An oral laxative for bowel cleansing (2 doses) the day before surgery.
  Drug: Metronidazole 1 g Intravenous An intravenous antibiotic pattern of metronidazole 1 g during anesthetic induction.
  Drug: Cefuroxime 1,5 g Intravenous An intravenous antibiotic pattern of cefuroxime 1,5 g during anesthetic induction.
  Interventions: Drug: Cefuroxime (750mg) I.V; Procedure: Colonic Surgery; Drug: Cefuroxime 750mg oral; Drug: Metronidazole 250 MG Oral Tablet [Flagyl]; Drug: Metronidazole 1 g Intravenous; Drug: Cefuroxime 1,5 g Intravenous; Drug: Sodium picosulfate, light magnesium oxide, anhydrous citric acid 10 mg/3.5 g/10.97 g Oral
- Oral + Parenteral prophylaxis (Active Comparator): Drug: Extra dosage - cefuroxime (750mg) I.V In both groups a second intravenous dose of cefuroxime (750mg) will be administered if the intraoperative time elongates more than three hours or there is an intraoperative bleeding over 1000cc
  Procedure: Colonic Surgery Both groups undergo colonic surgery. This section does not include rectal surgery ( see Inclusion/exclusion criteria)
  Drug: Cefuroxime 750mg oral An oral antibiotic pattern of ciprofloxacin (750mg / 12h, 2 doses) the day before surgery.
  Drug: Metronidazole 250mg oral An oral antibiotic pattern of metronidazole (250mg / 8h, 3 doses) the day before surgery.
  Drug: Metronidazole 1 gr Intravenous An intravenous antibiotic pattern of metronidazole 1 g during anesthetic induction.
  Drug: Cefuroxime 1,5 g Intravenous An intravenous antibiotic pattern of cefuroxime 1,5 g during anesthetic induction.
  Interventions: Drug: Cefuroxime (750mg) I.V; Procedure: Colonic Surgery; Drug: Cefuroxime 750mg oral; Drug: Metronidazole 250 MG Oral Tablet [Flagyl]; Drug: Metronidazole 1 g Intravenous; Drug: Cefuroxime 1,5 g Intravenous

INTERVENTIONS:
Drug: Cefuroxime (750mg) I.V — Extra dosage
Procedure: Colonic Surgery — Colonic Surgery
Drug: Cefuroxime 750mg oral — Oral prophylaxis
Drug: Metronidazole 250 MG Oral Tablet [Flagyl] — Oral prophylaxis
Drug: Metronidazole 1 g Intravenous — IV prophylaxis
Drug: Cefuroxime 1,5 g Intravenous — IV prophylaxis
Drug: Sodium picosulfate, light magnesium oxide, anhydrous citric acid 10 mg/3.5 g/10.97 g Oral — Laxative for bowel cleansing
  Arms: Oral + Parenteral prophylaxis + Mechanical Bowel Preparation

SUMMARY:
The ORALEV Study found that preoperative oral antibiotics can reduce the incidence of surgical site infections after colonic resection, compared with no preparation.

The role of mechanical bowel preparation in patients needing colonic surgery is yet to be elucidated.

No randomised controlled trials have assessed the impact of mechanical bowel preparation combined with oral antibiotics on the incidence of surgical site infections after colonic surgery, compared with oral antibiotics only.

DETAILED DESCRIPTION:
International, multicentre, pragmatic, parallel-group, randomised controlled trial.

Routine antibiotics for the intravenous and oral prophylaxis of colorectal surgery will be used.

Experimental group: Patients undergoing elective colonic surgery that involves colonic resection.

The antibiotic prophylaxis in this group will be composed of:

An oral antibiotic pattern of ciprofloxacin (750mg / 12h, 2 doses) and metronidazole (250mg / 8h, 3 doses) the day before surgery, plus mechanical bowel preparation with Sodium picosulfate, light magnesium oxide, and anhydrous citric acid (10 mg - 3.5 g - 10.97 g per dose/ 2 doses the day before surgery) + An intravenous antibiotics pattern of cefuroxime 1,5 g and metronidazole 1 g at anesthetic induction.

Control group: Patients undergoing elective colonic surgery that involves colonic resection.

The antibiotic prophylaxis in this group will be composed of:

An oral antibiotic pattern of ciprofloxacin (750mg / 12h, 2 doses) and metronidazole (250mg / 8h, 3 doses)

+ An intravenous antibiotic pattern of cefuroxime 1,5 g and metronidazole 1 gr at anesthetic induction.

In both groups a second intravenous dose of cefuroxime (750mg) will be administered if the intraoperative time prolongs for more than three hours or if there is an intraoperative bleeding over 1000cc.

There will not be a placebo treatment. Subject compliance will be evaluated according to the usual practice in surgical care field

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders, aged 18 years or above, with colonic disease without contraindications to surgical treatment, diagnosed with neoplasia or diverticular disease (diverticulosis with indication to elective surgery: stricture, chronic constipation), patients for whom a segmental or total colectomy is indicated.
* Patients who voluntarily accept to join the study and sign a dedicated written consent.
* Capability of understanding the study and take the medications prescribed.

Exclusion Criteria:

* Patients undergoing urgent surgery or no elective admission
* Patients who refuse to participate
* Patients with rectal disease or neoplasia
* Patients with pre-existing intrabdominal sepsis (abscess, acute diverticulitis)
* Patients who received preoperative antibiotic treatment for any other reasons during the two weeks before surgery
* Patients with Crohn's disease or ulcerative colitis
* Patients unlikely to adhere to the treatment prescribed
* Patients with allergy or contraindication to the medications used in the study
* Patients who need mechanical bowel preparation
* Patients with contraindication to bowel preparation used in the study (Citrafleet®):
* Patients with kidney failure needing haemodialysis or with hypermagnesemia
* Patients with severe heart failure
* Patients with gastric or duodenal ulcer
* Patients with mechanical obstruction
* Patients with toxic megacolon
* Patients with ascites or rhabdomyolysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 968 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Rate of Wound infection | 30 days
  Superficial, deep, body-cavity This is a Clinical measure supported by image if necessary All the morbidity problems are reported independently

SECONDARY OUTCOMES:
Local complications | 30 days after surgery
  Hematoma, seroma, evisceration
  This is a Clinical measure. This morbidity problems are reported independently as a YES/NO variable
Impaired healing | 30 days after surgery
  This is a Clinical measure always supported by image tests. This morbidity problems are reported independently as a YES/NO variable
Occlusive problems | 30 days from surgery
  Intestinal occlusion, Anastomotic stenosis, Postoperative ileus
Nephro-urinary complications | 30 days after surgery
  Acute urinary retention, Acute renal failure, cystitis, pyelonephritis ...
  This is a Clinical measure supported by more specific tests if necessary. This morbidity problems are reported independently as a YES/NO variable
Adverse events related to drugs (Harms) | 30 days after surgery
  Any adverse event related with the drug
  •This morbidity problems are reported independently as a YES/NO variable
Time to complete recovery | 30 days after surgery
  Interval between hospital admission and complete recovery ("can be discharged")
Length of Hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  Hospital stay since colorectal surgery is done
Iatrogenic problems | 30 days after surgery
  Injury to structures such as ureters, bowel loops artery / veins .
  •This morbidity problems are reported independently as a YES/NO variable
Bleeding problems | 30 days after surgery
  Hemoperitoneum, abdominal hematoma,anastomotic bleeding
  •This morbidity problems are reported independently as a YES/NO variable
Cardiac complications | 30 days after surgery
  Acute myocardial infarction, angor pectoris , atrial fibrillation, acute pulmonary edema
  This is a Clinical measure supported by more specific tests if necessary. This morbidity problems are reported independently as a YES/NO variable Cardiologist report will be required for including this items
Respiratory complications | 30 days after surgery
  Pneumonia, Atelectasia, Pulmonary embolism, ARDS
  This is a Clinical measure always supported by image . This morbidity problems are reported independently as a YES/NO variable
Neurological complications | 30 days after surgery
  Disorientation, cerebral vascular accident,
  This is a Clinical measure. This morbidity problems are reported independently as a YES/NO variable. Neurologist report will be required beyond disorientation.
Postoperative intestinal problems | 30 days after surgery
  Postoperative diarrhoea, nausea and vomiting
Readmission | 30 days after surgery
  Need to be readmitted after discharge
Reintervention | 30 days after surgery
  Need to be reoperated
Perioperative Hypovolemia | Intraoperative assessment
  Signs or symptoms of hypovolemia not related with bleeding, as assessed by the anesthetist at surgery
Patient satisfaction with preparation received | within the 30 days from surgery
  Patient satisfaction with the preparation receivced, assessed with a Verbal Rating Scale (VRS) from 1 (minimum satisfaction) to 10 (maximum satisfaction)
Death | 30 days after surgery
  Patient death for any cause and patient death in relation with treatment received
Anastomotic leak | 30 days after surgery
  clinical, radiological or intraoperatively detected abdominal or pelvic leak or collection

OTHER OUTCOMES:
Complications at 60 days of follow up | 60 days after surgery
  Complications and events will be recorded at 60-day follow-up, including:
  * Primary Outcome Measure, Outcome 1: Rate of Wound infection
  * Secondary Outcome Measures: Outcomes 2-6 / Outcomes 9-16 / Outcome 19
Complications at 5 years of follow up | 5 years after surgery
  Complications and events will be recorded at 5-year follow-up, including:
  * Primary Outcome Measure, Outcome 1: Rate of Wound infection
  * Secondary Outcome Measures: Outcomes 2-6 / Outcomes 9-16 / Outcome 19
  * Readmission related with infections, with culture and antibiogram.
  * In patients with cancer, the following variables will also be collected: Local recurrence / Systemic recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Eloy Espín-Basany, MD PhD, Study Chair — Hospital Universitario Valle de Hebron, Barcelona; Gianluca Pellino, MD, PhD, Study Director — Hospital Universitario Valle de Hebron, Barcelona; Alejandro Solís-Peña, MD, PhD, Study Director — Hospital Universitario Valle de Hebron, Barcelona
Locations (10):
- Jinling Hospital, Nanjing, China
- General University Hospital of Patras, Pátrai, Greece
- Humanitas Research Hospital, Rozzano, Italy
- Tomsk Oncological Hospital, Tomsk, Russia
- Spain (5):
  - Hospital General Universitario Vall d´Hebron, Barcelona, Barcelona, Spain
  - Hospital de Bellvitge, Barcelona, Hospitalet de Llobregat, Barcelona, Spain
  - Hospital Universitario Cruces, Cruces
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario Ramón y Cajal, Madrid
- Royal Marsden Hospital, Imperial College of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pellino G, Solis-Pena A, Kraft M, Huguet BM, Espin-Basany E. Preoperative oral antibiotics with versus without mechanical bowel preparation to reduce surgical site infections following colonic resection: Protocol for an international randomized controlled trial (ORALEV2). Colorectal Dis. 2021 Aug;23(8):2173-2181. doi: 10.1111/codi.15681. Epub 2021 May 12. PMID 33872448
- [Derived] Willis MA, Toews I, Soltau SL, Kalff JC, Meerpohl JJ, Vilz TO. Preoperative combined mechanical and oral antibiotic bowel preparation for preventing complications in elective colorectal surgery. Cochrane Database Syst Rev. 2023 Feb 7;2(2):CD014909. doi: 10.1002/14651858.CD014909.pub2. PMID 36748942
- [Derived] Koskenvuo L, Sallinen V. Preoperative oral antibiotics in colon surgery. Lancet Gastroenterol Hepatol. 2020 Sep;5(9):801-802. doi: 10.1016/S2468-1253(20)30203-X. No abstract available. PMID 32818460